CLINICAL TRIAL: NCT04959331
Title: Clinical Effectiveness and Bacteriological Eradication of Three Different Short-course Antibiotic Regimens and Single-dose Fosfomycin for Uncomplicated Lower Urinary Tract Infections in Adult Women.
Brief Title: Clinical Effectiveness and Bacteriological Eradication of 4 Short-course Antibiotics for Uncomplicated UTIs in Women.
Acronym: SCOUT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Balearic Islands Health Service (Ibsalut) (Other); Instituto de Investigación Sanitaria Aragón (Other); Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IJG-SCOUT-2021
Record Dates: First submitted 2021-07-05; First posted 2021-07-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-02

CONDITIONS: Urinary Tract Infections
Keywords: Urinary Tract Infections; Women; Patient Outcome Assessment; Bacteriological Eradication; Urinalysis; Anti-Bacterial Agents; Antimicrobial Resistance; Short Course; Primary Health Care
MeSH Terms: conditions — Urinary Tract Infections | interventions — Fosfomycin; Nitrofurantoin; Amdinocillin Pivoxil

STUDY DESIGN:
Intervention Model Description: 3 short-course antibiotic regimens and one-dose of fosfomycin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Short-course fosfomycin (Active Comparator): 3 g of fosfomycin once daily for two days (sachets)
  Interventions: Drug: Fosfomycin Trometamol Salt
- Short-course nitrofurantoin (Active Comparator): Five-day nitrofurantoin 100 mg t.i.d. (pills)
  Interventions: Drug: Nitrofurantoin
- Short-course pivmecillinam (Active Comparator): Three-day pivmecillinam 400 mg. t.i.d. (pills)
  Interventions: Drug: Pivmecillinam
- Single-dose fosfomycin (Active Comparator): Single 3 g dose of fosfomycin (sachet)
  Interventions: Drug: Fosfomycin Trometamol Salt

INTERVENTIONS:
Drug: Fosfomycin Trometamol Salt — Fosfomycin 3 g 2 sachets, taken orally, once daily for two days
  Other Names: Monurol
  Arms: Short-course fosfomycin
Drug: Nitrofurantoin — Nitrofurantoin 50 mg pills, taken orally, two pills/8 hours, for five days
  Other Names: Furantoin
  Arms: Short-course nitrofurantoin
Drug: Pivmecillinam — Pivmecillinam 400 mg pills. taken orally, one pill/8 hours, for three days
  Other Names: Selexid
  Arms: Short-course pivmecillinam
Drug: Fosfomycin Trometamol Salt — Fosfomycin 3 g one sachet, taken orally, for one day
  Other Names: Monurol
  Arms: Single-dose fosfomycin

SUMMARY:
Randomized clinical trial in which women aged 18 or older and with symptoms of uncomplicated lower urinary tract infection and a positive urine dipstick analysis will be randomized to one of the following four groups: 2-day 3 g fosfomycin o.d., 3-day pivmecillinam 400 mg. t.i.d, 5-day nitrofurantoin 100 mg t.i.d. or a single dose of 3 g of fosfomycin. Sample: 1,000 patients. Two co-primary endpoints are considered: clinical effectiveness at day 7 and bacteriological eradication at day 14. Follow-up visits are scheduled at days 7 (phone call), 14 and 28 for assessing evolution. Urine samples will be collected in the three on-site visits and urine cultures performed.

DETAILED DESCRIPTION:
Uncomplicated lower urinary tract infections (LUTI) represent a common problem in primary care. Resistance of uropathogens to common antibiotics has significantly increased in the last years. Current local guidelines recommend the use of a single 3 g dose of fosfomycin for these infections, but most general practitioners prefer short-course therapies to single-dose therapy. No study has compared head-to-head short course antimicrobial agents for uncomplicated LUTIs. Therefore, the aim of this randomized clinical trial is to compare three different short-course antibiotic therapies with single-dose fosfomycin for uncomplicated LUTIs in adult women. This will be a pragmatic, multicenter, parallel group, open randomized trial. Women aged 18 or older and with symptoms of uncomplicated LUTI and a positive urine dipstick analysis will be randomized to one of the following four groups: 2-day 3 g fosfomycin o.d., 3-day pivmecillinam 400 mg. t.i.d, 5-day nitrofurantoin 100 mg t.i.d. or a single dose of 3 g of fosfomycin. Sample: 1,000 patients. Two co-primary endpoints are considered: clinical effectiveness, defined as resolution of symptoms, answered by the patients at day 7, and bacteriological eradication (proportion of patients bacteriologically cured) at day 14. Patients will be given a symptom diary for seven days. Follow-up visits are scheduled at days 7 (phone call), 14 and 28 for assessing evolution. Urine samples will be collected in the three on-site visits and urine cultures performed. If positive, antibiograms for the 3 antibiotics studied will be performed.

ELIGIBILITY:
Inclusion Criteria:

Women of 18 years of age or older, with clinical features of uncomplicated community-acquired lower urinary tract infection including:

* At least one of four key symptoms of lower urinary tract infection: dysuria, urgency including nycturia, frequency, and suprapubic tenderness that could be attributed to an uncomplicated lower urinary tract infection, and no alternative explanation (i.e. symptoms suggestive of sexually-transmitted infection or vulvovaginitis), and
* A urine dipstick analysis positive for either nitrites or leukocyte esterase.

Exclusion Criteria:

* Male sex
* High suspicion of pyelonephritis (i.e. fever ≥ 37.5°C or flank pain/tenderness)
* Any condition that may lead or predispose to complicated urinary infection (i.e. indwelling urinary catheter, pregnancy, immunosuppressive therapy, abnormal urinary tracts, recurrent urinary tract infection, severe neurological disease affecting the bladder)
* Pregnancy or planned pregnancy
* Symptoms consistent with urinary tract infection in the preceding 4 weeks
* Patients taking long-term antibiotic prophylaxis
* Ongoing antibiotic therapy or use of any systemic antibiotic in the previous 7 days
* Symptoms correlating with differential diagnosis (i.e. vaginal discharge or pain)
* Hypersensitivity or allergy to β lactams, nitrofurantoin and/or fosfomycin
* Moderate to severe chronic renal insufficiency
* Pre-existing polyneuropathy
* History of lung or liver reaction or peripheral neuropathy after previous use of nitrofurantoin
* Glucose-6-phosphate dehydrogenase deficiency
* Porphyria or systemic primary carnitine deficiency or of the type organic aciduria (i.e. methylmalonic aciduria and propionicacidaemia)
* Esophageal stricture
* Current intake of allopurinol or probenecid or valproate
* Currently part of another randomized clinical trial
* Previous enrolment in the proposed study
* Patients living in long-term institutions; and/or
* Difficulty in conducting scheduled follow-up visits

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical effectiveness. | Day 7.
  Proportion of patients who report being cured, defined as the resolution of the four symptoms, scoring 0 in the symptom diary.
Bacteriological eradication. | Day 14.
  Proportion of patients bacteriologically cured, defined as less than 1,000 colony forming units (cfu)/ml.

SECONDARY OUTCOMES:
Duration of symptoms. | From baseline visit to day 7.
  Number of days until the last day the patient scores 0 in any of the four symptoms.
Bacteriological eradication. | Day 28.
  Proportion of patients bacteriologically cured, defined as less than 1,000 cfu/ml.
Relapse rate. | Days 7, 14 and 28.
  Proportion of patients presenting a relapse of symptoms within the first four weeks after inclusion in the study and timing of relapse of symptoms and/or bacteriuria.
Reattendance and complication rate. | Days 7, 14 and 28.
  Proportion of patients re-attending healthcare services and development of complications within the first 4 weeks (i.e. pyelonephritis, urosepsis).
Adverse event rate. | Days 7, 14 and 28.
  Proportion of patients presenting adverse and serious adverse events.
Change in quality of life. | Days 0 and 7.
  Change in the quality of life by means of the 5-level EQ-5D version (EQ-5D-5L) validated questionnaire (Spanish version).

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Morros, MD PhD, Study Chair — Pharmacist
Locations (33):
- Spain (33):
  - Calatayud Center, Calatayud, Aragon
  - Las Fuentes Center, Zaragoza, Aragon
  - Arrabal Health Center, Zaragoza, Aragon
  - Parque Goya Health Center, Zaragoza, Aragon
  - Santa Ponça Health Center, Calvià, Balearic Islands
  - Emili Darder Center, Palma de Mallorca, Balearic Islands
  - Camp Redó Health Center, Palma de Mallorca, Balearic Islands
  - Son Pisà Center, Palma de Mallorca, Balearic Islands
  - Son Serra-La Vileta Health Center, Palma de Mallorca, Balearic Islands
  - Santa Maria del Camí Center, Santa Maria del Camí, Balearic Islands
  - Banyoles Center, Banyoles, Catalonia
  - Corbera Center, Corbera de Llobregat, Catalonia
  - La Gavarra Health Center, Cornellà de Llobregat, Catalonia
  - 17 de Setembre Center, el Prat de Llobregat, Catalonia
  - Can Vidalet Center, Esplugues de Llobregat, Catalonia
  - Santa Clara Center, Girona, Catalonia
  - Florida Center, L'Hospitalet de Llobregat, Catalonia
  - Can Serra Center, L'Hospitalet de Llobregat, Catalonia
  - Montblanc Center, Montblanc, Catalonia
  - Pere Garau Center, Palma de Mallorca, Catalonia
  - Molí Nou Center, Sant Boi de Llobregat, Catalonia
  - Sant Feliu de Guíxols Center, Sant Feliu de Guíxols, Catalonia
  - Sant Just Desvern Center, Sant Just Desvern, Catalonia
  - Vila Vella Center, Sant Vicenç dels Horts, Catalonia
  - Jaume I Health Center, Tarragona, Catalonia
  - El Puerto Center, Coslada, Madrid
  - Valleaguado Health Center, Coslada, Madrid
  - Los Alpes Health Center, Madrid, Madrid
  - Aquitania Health Center, Madrid, Madrid
  - Mar Báltico Center, Madrid, Madrid
  - Buenos Aires Center, Madrid, Madrid
  - San Fernando Health Center, San Fernando de Henares, Madrid
  - Villarejo de Salvanés Health Center, Villarejo de Salvanés, Madrid

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: On request after publication.
Access Criteria: Principal investigator's email (carles.llor@gmail.com)

REFERENCES:
- [Derived] Garcia-Sangenis A, Morros R, Aguilar-Sanchez M, Medina-Perucha L, Leiva A, Ripoll J, Martinez-Pecharroman M, Bartolome-Moreno CB, Magallon Botaya R, Marin-Canada J, Molero JM, Moragas A, Troncoso A, Monfa R, Llor C; SCOUT Study Group. Clinical effectiveness and bacteriological eradication of three different Short-COurse antibiotic regimens and single-dose fosfomycin for uncomplicated lower Urinary Tract infections in adult women (SCOUT study): study protocol for a randomised clinical trial. BMJ Open. 2021 Nov 25;11(11):e055898. doi: 10.1136/bmjopen-2021-055898. PMID 34824124